CLINICAL TRIAL: NCT01556906
Title: A Phase II Open Label, Dose-Escalation Study to Determine the Safety, Tolerability and Efficacy of Microsomal Triglyceride Transfer Protein (MTP) Inhibitor BMS-201038 in Patients With Homozygous Familial Hypercholeterolemia
Brief Title: Safety, Tolerability and Efficacy of Microsomal Triglyceride Protein (MTP) Inhibitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Collaborators: University of Pennsylvania (Other); Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP1001
Record Dates: First submitted 2012-03-07; First posted 2012-03-19 (Estimated); Results first posted 2013-02-22 (Estimated); Last update posted 2013-04-10 (Estimated); Status verified 2013-04

CONDITIONS: Homozygous Familial Hypercholesterolemia
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — BMS201038

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lomitapide (Experimental): This is an open label trial where all patients receive lomitapide (AEGR733/BMS-201038)at escalating doses
  Interventions: Drug: Lomitapide

INTERVENTIONS:
Drug: Lomitapide — Oral administration with escalating doses administered once daily
  Other Names: AEGR-733; BMS-201038

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of 4 doses of lomitapide (AEGR-733; BMS-201038) given as an initial low dose and then escalated through an additional 3 dose levels over a 16-week period.

The secondary objectives of this study included the evaluation of the pharmacodynamics of lomitapide based on:

* Percent change in low-density lipoprotein cholesterol (LDL-C), total cholesterol (TC), triglycerides, and very low density lipoprotein cholesterol (VLDL-C) concentrations at the end of each 4-week dosing period compared to the Baseline value of each parameter at the end of the previous dose phase(s).
* Changes in other plasma lipoproteins: apolipoproteins (apo B, apo AI, apo AII, apo CIII, apo E) and lipoprotein a [Lp(a)].

DETAILED DESCRIPTION:
This is a single center, open-label, Phase 2 clinical trial designed to evaluate the safety, tolerability, and pharmacodynamics of lomitapide in the treatment of patients with homozygous familial hypercholesterolemia (HoFH).

Patients are required to stop all lipid-lowering therapies, including apheresis, within 4 weeks prior to the Baseline visit and throughout the study. Patients are placed on a rigorous low-fat diet (<10% of energy from total dietary fat) at the Screening assessment; dietary counseling by a registered dietitian will be initiated at Screening and will continue at each subsequent study visit.

Patients initially receive 0.03 mg/kg of lomitapide orally every day for 4 weeks. Intra-patient dose escalation to 0.1 mg/kg, 0.3 mg/kg/day and 1.0 mg/kg/day occur every 4 weeks if specific protocol-defined stopping rules related to Grade 3 or 4 toxicities or serious adverse events (SAEs) do not apply.

The study includes 15 study visits over 22 weeks: a Screening visit (Visit 1) conducted within 2 weeks prior to dosing, a Baseline visit (Visit 2) conducted on Day 1 prior to the first dose, 12 visits conducted during the treatment period (Visits 3 through 14), and a Follow-up visit (Visit 15) conducted approximately 4 weeks after the last dose of lomitapide.

Screening and Baseline procedures include medical and medication history, physical examination, vital signs, 12-lead electrocardiogram (ECG), pulmonary function tests (PFTs), safety laboratory tests, fat soluble vitamin levels and a fatty acid profile. Nuclear magnetic resonance spectroscopy (NMRS) of the liver will be conducted at Baseline, at the end of each dosing period, and at the follow up visit to assess hepatic fat content. Baseline efficacy assessment includes a fasting lipid profile (TC, LDL-C [directly measured], VLDL-C, high density lipoprotein-cholesterol [HDL-C], triglycerides, and apolipoproteins [apo B, apo AI, apo AII, apo CIII, apo E] and Lp(a)).

Safety and lipid profile assessments are repeated during the treatment period and at the Follow-up visit conducted 28 days after the last dose of lomitapide.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥13 years of age
2. Clinical diagnosis of HoFH AND one of the following (a, b, or c):

   * Documented functional mutation in both LDL receptor alleles, OR
   * Skin fibroblast LDL receptor activity <20% of normal, OR
   * TC >500 mg/dL AND triglycerides < 300 mg/dL AND both parents with documented TC >250 mg/dL
3. Body weight ≥40 kg
4. Negative screening pregnancy test if female of child-bearing potential
5. Subjects must be willing and able to comply with all study-related procedures
6. Subjects must be willing and able to go off all lipid-lowering medications, dietary supplements (psyllium preparations) and LDL apheresis within 4 weeks prior to the Baseline visit until the end of the study.

Exclusion Criteria:

1. Uncontrolled hypertension defined as: systolic blood pressure >180 mmHg, diastolic blood pressure >95 mmHg
2. History of chronic renal insufficiency (serum creatinine >2.5 mg/dL)
3. History of liver disease or abnormal LFTs at screening (>3x upper limit of normal [ULN])
4. Any major surgical procedure occurring < 3 months prior to the screening visit
5. Cardiac insufficiency defined by the New York Heart Association classification as functional Class III or Class IV
6. History of a non-skin malignancy within the previous 5 years
7. History of alcohol or drug abuse
8. Participation in an investigational drug study within 6 weeks prior to the screening visit
9. Serious or unstable medical or psychological conditions that, in the opinion of the Investigator, would compromise the patient's safety or successful participation in the study.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2003-06; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan J Rader, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Cuchel M, Bloedon LT, Szapary PO, Kolansky DM, Wolfe ML, Sarkis A, Millar JS, Ikewaki K, Siegelman ES, Gregg RE, Rader DJ. Inhibition of microsomal triglyceride transfer protein in familial hypercholesterolemia. N Engl J Med. 2007 Jan 11;356(2):148-56. doi: 10.1056/NEJMoa061189. PMID 17215532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed from 05 Jun 2003 to 16 Feb 2004. The study was performed at a single medical clinic.
Groups:
- Lomitapide Escalated: Lomitapide initiated with an oral dose of 0.03 mg/kg/day for 4 weeks and then escalated through an additional 3 dose levels (0.1, 0.3, and 1.0 mg/kg/day) every 4 weeks over a 16-week period.
Period: Overall Study
Arm/Group | Lomitapide Escalated
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
Age Continuous [Mean (Standard Deviation); unit: years] | 25.7 (9.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: LDL-C
Description: Percent change in LDL-C compared to Baseline.
Time Frame: Up to 16 weeks of treatment comapred to Baseline
Population: All patients treated
Measure: Mean (Standard Deviation); unit: percentage change in LDL-C
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
percentage change in LDL-C | -50.94 (9.311)

2. Secondary Outcome: Absolute Change From Baseline in Alanine Aminotransferase (ALT)
Description: Absolute change from Baseline in ALT
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
U/L | 91.2 (85.53)

3. Secondary Outcome: Absolute Change From Baseline in Aspartate Aminotransferase (AST)
Description: Absolute change from Baseline in AST
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
U/L | 37.5 (32.51)

4. Secondary Outcome: Absolute Change From Baseline in Total Bilirubin
Description: Absolute change from Baseline in total bilirubin
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
mg/dL | -0.25 (0.274)

5. Secondary Outcome: Absolute Change From Baseline in Hepatic Fat Percent
Description: Absolute change from Baseline in hepatic fat percent
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: percent of hapatic fat
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
percent of hapatic fat | 19.3 (12.92)

6. Secondary Outcome: Absolute Change From Baseline in Forced Expiratory Volume During 1 Second (FEV1)
Description: Absolute change from Baseline in FEV1
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
Liters | 0.070 (0.2406)

7. Secondary Outcome: Absolute Change From Baseline in Carbon Monoxide Lung Diffusing Capacity (DLCO)(a Pulmonary Function Test)
Description: Absolute change from Baseline in DLCO
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mL CO/min/mm Hg
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
mL CO/min/mm Hg | -3.020 (5.3246)

8. Secondary Outcome: Absolute Change From Baseline in Vitamin A
Description: Absolute change from Baseline in vitamin A
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
µmol/L | -0.35 (0.847)

9. Secondary Outcome: Absolute Change From Baseline in Vitamin E
Description: Absolute change from Baseline in vitamin E
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
umol/L | -94.35 (130.797)

10. Secondary Outcome: Absolute Change From Baseline in Vitamin D
Description: Absolute Change From Baseline in Vitamin D
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
nmol/L | -6.57 (10.712)

11. Secondary Outcome: Absolute Change From Baseline in Ratio of Vitamin E to Total Lipids
Description: Absolute Change From Baseline in ratio of vitamin E to total lipids
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
ratio | -0.0 (1.71)

12. Secondary Outcome: Absolute Change From Baseline in Alpha Linoleic Acid (ALA)
Description: Absolute Change From Baseline in ALA
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
mg/mL | 0.06 (0.045)

13. Secondary Outcome: Absolute Change From Baseline in Eicosapentaenoic Acid (EPA)
Description: Absolute Change From Baseline in EPA
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
mg/mL | -0.08 (0.079)

14. Secondary Outcome: Absolute Change From Baseline in Docosahexaenoic Acid (DHA)
Description: Absolute Change From Baseline in DHA
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
mg/mL | -0.08 (0.045)

15. Secondary Outcome: Absolute Change From Baseline in Linoleic Acid (LA)
Description: Absolute Change From Baseline in LA
Time Frame: Baseline and 16 weeks of treatment
Population: All patients treated
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Lomitapide Escalated
Number analyzed (Participants) | 6
mg/mL | -2.9 (1.51)

ADVERSE EVENTS:
Time Frame: First dose through 28 days post-treatment
Arm/Group | Lomitapide Escalated
Serious Adverse Events (participants affected / at risk) | 1/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lomitapide Escalated (N=6)
Breast mass (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lomitapide Escalated (N=6)
Diarrhoea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Alinine aminotransferase increased (Investigations) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 3
Aspartate aminotransferase increased (Investigations) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dizziness (Nervous system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hot flush (Vascular disorders) | 1
International normalized ratio increased (Investigations) | 2
Asthenia (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Scratch (Injury, poisoning and procedural complications) | 1
Xanthoma (Skin and subcutaneous tissue disorders) | 1
Eye disorders (Eye disorders) | 1
Rhinitis (Infections and infestations) | 1
Prothrombin time prolonged (Investigations) | 1
Breast mass (Reproductive system and breast disorders) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Chest pain (General disorders) | 1
Haemoglobinuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Information is unavailable.